CLINICAL TRIAL: NCT04045496
Title: A Phase 1, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-3312 in Adult Patients With Advanced Solid Tumors
Brief Title: A First-in-Human, Phase 1 Study of JAB-3312 in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAB-3312-1001
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer; Colorectal Cancer; Pancreatic Ductal Carcinoma; Esophageal Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma; Breast Cancer; Other Solid Tumors
Keywords: Src homology phosphatase 2 (SHP2); PTPN11; Kirsten rat sarcoma (KRAS) proto-oncogene, GTPase; epidermal growth factor receptor (EGFR)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Carcinoma, Pancreatic Ductal; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Noonan Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JAB-3312 (Experimental): JAB-3312 will be administered orally once daily in 21 days treatment cycles.
  Interventions: Drug: JAB-3312

INTERVENTIONS:
Drug: JAB-3312 — JAB-3312 will be supplied as 0.25 mg and 1.0 mg capsules.

SUMMARY:
This is a Phase 1, first-in-human, open-label dose-escalation study to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) and assess the DLT of JAB-3312. It is anticipated that approximately 24 subjects will be enrolled in the dose-escalation phase of the study. JAB-3312 will be administered orally once daily (QD) in 21-day treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥18 years-of-age at the time of signature of the informed consent form (ICF).
2. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
3. Subjects with histologically or cytologically confirmed advanced solid tumors which have progressed despite standard therapy or for which no standard therapy exists.
4. Subjects with life expectancy ≥3 months.
5. Patients must have at least one measurable lesion as defined by RECIST v1.1.
6. Patients who have sufficient baseline organ function.

Exclusion Criteria:

1. Severe autoimmune disease (including immune-related adverse events of prior immune-oncology therapy) or autoimmune disorder that requires chronic systemic corticosteroid treatment at immunosuppressive doses (prednisone >10 mg/day or equivalent).
2. Known malignant central nervous system disease other than neurologically stable, treated brain metastases.
3. History or evidence of interstitial lung disease, radiation pneumonitis which required steroid treatment, or idiopathic pulmonary fibrosis, pleural or pericardial effusion that required intervention such as a drain.
4. 8. History of seropositive status for hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
5. History or evidence of active infections (Grade ≥2).
6. History or evidence of significant inflammatory or vascular eye disorder.
7. History of an allogeneic bone marrow or solid organ transplant.
8. Use of systemic anti-cancer agent (except for anti-androgen therapy for prostate cancer) or investigational drug ≤28 days prior to the first dose of JAB-3312.
9. History of radiation therapy ≤28 days prior to the first dose of JAB-3312, or likely to require radiation therapy at any time until the 30 days after the last dose of JAB-3312.
10. History of transfusion of whole blood, red blood cell or platelet packets ≤2 weeks before the start of treatment.
11. Subjects experiencing unresolved Grade >1 toxicity before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | Approximately 2 years
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle with JAB-3312.
Find Recommended Phase 2 Dose (RP2D) of JAB-3312 | Approximately 2 years
  Measurements of MTD (i.e. the highest dose of JAB-3312 associated with the occurrence of Dose Limiting Toxicities (DLTs) in <33% of patients) or the RP2D (i.e. the highest tested dose that is declared safe and tolerable by the Investigators and Sponsor)

SECONDARY OUTCOMES:
Number of participants with adverse events | Approximately 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments
Area under the curve | Approximately 2 years
  Area under the plasma concentration time curve of JAB-3312
Cmax | Approximately 2 years
  Highest observed plasma concentration of JAB-3312
Tmax | Approximately 2 years
  Time of highest observed plasma concentration of JAB-3312
T1/2 | Approximately 2 years
  Half life of JAB-3312
Objective response rate ( ORR ) | Approximately 2 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
Duration of response ( DOR ) | Approximately 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobio Pharmaceuticals, Study Director — Jacobio Pharmaceuticals
Locations (4):
- United States (4):
  - HealthONE Clinic Services Oncology-Hematology, Denver, Colorado
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Washington University School of Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No